CLINICAL TRIAL: NCT04942470
Title: Phd Candidate/Specialist Surgery Nurse
Brief Title: Effect of Aloe Vera and Propolis on Wound Healing in Pressure Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Özgül Aydemir, PHD Candidate, Surgery Specialist Nurse, Haydarpasa Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OAydemir1673348861.; PHD Candidate (Registry Identifier: İSTANBUL UNIVERSITY-CERRAHPAŞA)
Record Dates: First submitted 2021-04-21; First posted 2021-06-28 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Pressure Ulcer
Keywords: Aloe Vera; Propolis; Pressure ulcer prevention; Nursing care; Treatment
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: The research was planned as an experimental study with a randomized control group to determine the effect of Aloe Vera and Propolis on wound healing in pressure injuries.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental:Intervention Arm (Experimental): For the experimental group patients, sponges prepared by impregnating cream containing Aloe Vera and Propolis will be sterilized in the sterilization device. If any contamination occurs in the wound area of the patient (in the presence of feces, discharge), the product is applied to the wound bed after cleaning the wound with 0.9% isotonic sodium chloride washing solution. And the effects of the product on the wound will be monitored. The solution will be applied 2 times a day for the first 10 days. The second 10 days will be applied daily 1x1. Application results will be recorded and wound healing status will be monitored. In order to prevent and maintain pressure injury, the experimental group patients will be given an in-bed position every 2 hours. If there is a deficiency or deterioration in the patient's laboratory findings (hemoglobin, albumin, prealbumin, leukocyte, blood sugar, SaO2, fever, pulse, blood pressure, etc.), necessary treatment and care is performed.
  Interventions: Other: Aloe vera and propolis applied
- No Intervention:Control Arm (No Intervention): In control group patients, if any pollution occurs in the wound area (feces, discharge) in the sterile dressing performed in the morning and evening at 10-22 hours, the wound area will be cleaned with the help of 0.9% isotonic sodium chloride washing solution and the clinical routine application of the pressure injury of the hospital will be carried out according to the physician's order. In patients in the control group, the results of the application will be recorded and wound healing status will be observed. An in-bed position will be given every 2 hours for the prevention and care of pressure injury patients of the control group patients. If there is a deficiency or deterioration in the patient's laboratory findings (hemoglobin, albumin, prealbumin, leukocyte, blood sugar, SaO2, fever, pulse, blood pressure and other), the necessary treatment and care will be performed.

INTERVENTIONS:
Other: Aloe vera and propolis applied — Suitable of sterile pads containing aloe vera and propolis to the area with pressure sores
  Arms: Experimental:Intervention Arm

SUMMARY:
This study was planned as an experimental study with a randomized control group to determine the effect of Aloe Vera and Propolis on wound healing in pressure injuries.

After receiving ethical approval, this study will take place between January 30, 2021 and January 30, 2022 in the General Intensive Care Unit of The Haydarpasa Numune Training and Research Hospital of the Istanbul Provincial Health Directorate, according to the criteria for inclusion and exclusion. The purpose of the research will be explained and it will be selected in accordance with the research criteria from individuals in the universe who have been granted permission by themselves or their guardians to participate in the post-information research. Within the scope of the planned study, an academic study containing aloe vera and propolis cream for patients with pressure injury and reporting the sample size to be used to determine the effect of the solution prepared by the researcher on wound healing (1) In the light of study , standard deviations for groups, respectively, in order to find a statistical difference of 20.4 days (50.5 days) from the 63.2 ± taken as the average wound healing time in pressure injuries; If 20,4 and 15 are taken, the effective sample size calculated for double-sided Student's t test for 0.05 error level and minimum 80% power is calculated as 33 for each group and a total of 66 patients will be admitted to the trial and control group. Patients who meet the study criteria will be distributed daily to experimental and control groups through a computerized randomization program.After randomization, in order to collect data, developed by the researcher in line with the relevant literature information; 'Patient Diagnostic Form', 'Braden Pressure Injury Risk Assessment Scale', 'Bates-Jensen Wound Assessment Tool' and 'Wound Surface 3D Assessment System (Ekare/inSight®)' will be used for wound measurement.In the collection of the data of the patients in the experimental and control group, the patient will be accepted according to the criteria of inclusion and exclusion in the research. 'Patient Diagnostic Form', 'Health History', 'Patient Measurements (Life Findings and Laboratory Findings)' will be questioned and recorded in the experimental and control group patients. The total scores of the test group patients will be recorded by performing a risk assessment with the pressure wound, 'Braden Pressure Injury Risk Assessment Scale'. With the 'Bates-Jensen Wound Assessment Tool', the physiological characteristics of the wound and the condition of the wound will be measured and recorded by performing wound staging. With ekare/inSight® device, wound staging will be performed by photographing the wound area, at the same time the healing status of the wound will be monitored and the reduction in wound volume, i.e. healing, will be observed. With ekare/inSight® device, the healing stages of the wound will be recorded. In the 'Braden Pressure Injury Risk Scale Assessment', the scores and total scores of the patients in the 'Braden Pressure Injury Risk Scale Assessment' will be recorded on the one day, the fourth day, the seventh day, the fourteenth day and twenty-first days by evaluating the substances 'emotional perception', 'humidity', 'activity', 'mobilization', 'nutrition', 'friction/tearing'. Pressure injury risk status and recovery status of the test and control group patients will be measured by Bates-Jensen scores and Braden scores and evaluated on the one day, fourth day, seventh day, fourteen days and twenty-first days. In addition, the date of the wound culture and wound culture results will be recorded as the wound healing time of the patients in the experimental and control group.

DETAILED DESCRIPTION:
This research was planned as a randomized controlled experimental research to determine the effect of Aloe Vera and Propolis on wound healing in pressure injuries.

According to the European Pressure Injuries Advisory Panel (EPUAP) definition, pressure injuries alone are localized skin and/or subsurned tissue damage caused by pressure by pressure or tearing, usually occuring on bone protrusions (2).

Pressure injuries that we often encounter in the intensive care unit cause significant problems such as pain and discomfort, low movement and addiction in patients, increased mortality and morbidity, as well as a significant increase in the cost of health care in addition to loss of work and time (1).

Despite recent advances in wound care products, traditional treatments based on naturally sourced compounds such as plant extracts, honey and larvae remain important as alternative treatment options today. Today's trend is more towards the development of innovative wound care treatments, combining the use of traditional healing agents and modern products/applications.

In one study, they developed a transparent treatment by adding aloe vera to alginate hydrogels, propolis to dressing films, and layers of hydrogel containing honey (3). Studies have found that Aloe vera has an effect on the wound healing process as well as its antioxidant, antibacterial, antifungal, antiviral, and immunomodulatory effects. Anti-inflammatory and antimicrobial activities; It facilitates wound healing by stimulating cell proliferation, collagen synthesis and angiogenesis and accelerating wound contraction (3;4).

In the literature, it is mentioned that propolis has antioxidant, anti-inflammatory and antibacterial activity on wound healing within alternative treatment methods.

In a study conducted on experimental animals titled "Wound Healing Activity of Western Algerian Propolis", they formed three groups. In this study where the treatment period was 23 days, the percentage of wound closure was 94.93 ± 5.29% in the first group where propolis was applied, 79.97 ± 13.01% in the second group where a commercial cream was applied, and 72.55 ± 19.94% in the third group without any application. In addition, it was observed that the wound healed in 12 days in the first group, 16 days in the second group and 18 days in the third group. As a result of this study, it was found that the rate of recovery was higher and faster in the group treated with propolis (5).

In addition to studies examining the effectiveness of aloe vera and propolis separately on wound healing, in a study in which they were applied together, their study on 'Medicinal Plant Extracts and the Use of Wound Closure Substances', active ingredients of various herbs such as Propolis and Aloe vera in wound healing and tissue regeneration reported that it can be used to induce the process of wound closure and thus reduce the time to complete wound closure (7). In addition, it is stated in various studies and literature that Aloe vera and propolis may be effective in pressure injuries, which are of great importance in chronic wounds (3; 6; 7).

This study will set an example for pressure injuries with chronic wounds, speeding up the healing time of the patient's wound area, early discharge, reducing maintenance costs and other studies.In the light of these resources, the approval of the institution was obtained from the Istanbul Provincial Health Directorate and pilot work was started on 11.03.2021. Patients were randomized and the data collection phase started.

ELIGIBILITY:
Inclusion Criteria:

* To agree verbally and in writing to participate in the research by himself or his legal guardian after the information for the research,
* Being 18 years of age or older,
* During the pressure wound stages of the participant in the study; Patients with stage II-III pressure sores
* The patients with iskial, sacral, thoracenthers, shoulder, dorsal, heel, malleos, pretibial, elbows, scapula, occiputal, the other regions that may form pressure injury to the body will be included in the study.

Exclusion Criteria:

* Those who have an allergic reaction to the solution to be applied,
* Individuals under the age of 18,
* Patients with Stage Ive IV pressure sores,
* If the patient is included in the study, it will be left out of the study if it loses life during the twenty-day period.
* Patients who do not agree to participate in the research verbally and in writing by themselves or their legal guardian after the information for the research will be excluded from the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-06-11 (Actual)

PRIMARY OUTCOMES:
Braden Pressure Injury Risk Scale Assessment | Day one scores
  Braden Pressure Injury Risk Scale Assessment
Braden Pressure Injury Risk Scale Assessment | Fourth day scores
  Braden Pressure Injury Risk Scale Assessment
Braden Pressure Injury Risk Scale Assessment | Seventh day scores
  Braden Pressure Injury Risk Scale Assessment
Braden Pressure Injury Risk Scale Assessment | Fourteenth day scores
  Braden Pressure Injury Risk Scale Assessment
Braden Pressure Injury Risk Scale Assessment | Twenty-first day scores
  Braden Pressure Injury Risk Scale Assessment
Bates-Jensen Wound Assessment Tool Scores | Day one scores
  Bates-Jensen Wound Assessment Tool Scores
Bates-Jensen Wound Assessment Tool Scores | Fourth day scores
  Bates-Jensen Wound Assessment Tool Scores
Bates-Jensen Wound Assessment Tool Scores | Seventh day scores
  Bates-Jensen Wound Assessment Tool Scores
Bates-Jensen Wound Assessment Tool Scores | Fourteenth day scores
  Bates-Jensen Wound Assessment Tool Scores
Bates-Jensen Wound Assessment Tool Scores | Twenty-first day scores
  Bates-Jensen Wound Assessment Tool Scores
Patient Measurements (Life Findings, Laboratory Values) | Day one hemoglobin measurement results (g/dL)
  Hemoglobin measurement results (g/dL)
Patient Measurements (Life Findings, Laboratory Values) | Fourth day hemoglobin measurement results (g/dL)
  Hemoglobin measurement results (g/dL)
Patient Measurements (Life Findings, Laboratory Values) | Seventh day hemoglobin measurement results (g/dL)
  Hemoglobin measurement results (g/dL)
Patient Measurements (Life Findings, Laboratory Values) | Fourteenth day hemoglobin measurement results (g/dL)
  Hemoglobin measurement results (g/dL)
Patient Measurements (Life Findings, Laboratory Values) | Twenty-first day hemoglobin measurement results (g/dL)
  Hemoglobin measurement results (g/dL)
Patient Measurements (Life Findings, Laboratory Values) | Day one albumın measurement results (g/dL)
  Albumın measurement results (g/dL)
Patient Measurements (Life Findings, Laboratory Values) | Seventh day albumın measurement results (g/dL)
  Albumın measurement results (g/dL)
Patient Measurements (Life Findings, Laboratory Values) | Fourteenth day albumın measurement results (g/dL)
  Albumın measurement results (g/dL)
Patient Measurements (Life Findings, Laboratory Values) | Twenty-first day albumın measurement results (g/dL)
  Albumın measurement results (g/dL)
Patient Measurements (Life Findings, Laboratory Values) | Day one pre-albumin measurement results (g/dL)
  Pre-albumin measurement results (g/dL)
Patient Measurements (Life Findings, Laboratory Values) | Seventh day pre-albumin measurement results (g/dL)
  Pre-albumin measurement results (g/dL)
Patient Measurements (Life Findings, Laboratory Values) | Fourteenth day pre-albumin measurement results (g/dL)
  Pre-albumin measurement results (g/dL)
Patient Measurements (Life Findings, Laboratory Values) | Twenty-first day pre-albumın measurement results (g/dL)
  Pre-albumin measurement results (g/dL)
Patient Measurements (Life Findings, Laboratory Values) | Day one glucose measurement results (mg/dL)
  Glucose measurement results (mg/dL)
Patient Measurements (Life Findings, Laboratory Values) | Fourth day glucose measurement results (mg/dL)
  Glucose measurement results (mg/dL)
Patient Measurements (Life Findings, Laboratory Values) | Seventh day glucose measurement results (mg/dL)
  Glucose measurement results (mg/dL)
Patient Measurements (Life Findings, Laboratory Values) | Fourteenth day glucose measurement results (mg/dL)
  Glucose measurement results (mg/dL)
Patient Measurements (Life Findings, Laboratory Values) | Twenty-first day glucose measurement results (mg/dL)
  Glucose measurement results (mg/dL)
Patient Measurements (Life Findings, Laboratory Values) | Day one leukocyte measurement results (10^3/uL)
  Leukocyte measurement results (10^3/uL)
Patient Measurements (Life Findings, Laboratory Values) | Fourth day leukocyte measurement results (10^3/uL)
  Leukocyte measurement results (10^3/uL)
Patient Measurements (Life Findings, Laboratory Values) | Seventh day leukocyte measurement results (10^3/uL)
  Leukocyte measurement results (10^3/uL)
Patient Measurements (Life Findings, Laboratory Values) | Fourteenth day leukocyte measurement results (10^3/uL)
  Leukocyte measurement results (10^3/uL)
Patient Measurements (Life Findings, Laboratory Values) | Twenty-first day leukocyte measurement results (10^3/uL)
  Leukocyte measurement results (10^3/uL)
Patient Measurements (Life Findings, Laboratory Values) | Day one SaO2 measurement results (%)
  SaO2 measurement results (%)
Patient Measurements (Life Findings, Laboratory Values) | Fourth day SaO2 measurement results (%)
  SaO2 measurement results (%)
Patient Measurements (Life Findings, Laboratory Values) | Seventh day SaO2 measurement results (%)
  SaO2 measurement results (%)
Patient Measurements (Life Findings, Laboratory Values) | Fourteenth day SaO2 measurement results (%)
  SaO2 measurement results (%)
Patient Measurements (Life Findings, Laboratory Values) | Twenty-first day SaO2 measurement results (%)
  SaO2 measurement results (%)
Patient Measurements (Life Findings, Laboratory Values) | Day one body temperature measurement results (degrees centigrade)
  Body Temperature measurement results (degrees centigrade)
Patient Measurements (Life Findings, Laboratory Values) | Fourth day body temperature measurement results (degrees centigrade)
  Body Temperature measurement results (degrees centigrade)
Patient Measurements (Life Findings, Laboratory Values) | Seventh day body temperature measurement results (degrees centigrade)
  Body Temperature measurement results (degrees centigrade)
Patient Measurements (Life Findings, Laboratory Values) | Fourteenth day body temperature measurement results (degrees centigrade)
  Body Temperature measurement results (degrees centigrade)
Patient Measurements (Life Findings, Laboratory Values) | Twenty-first day body temperature measurement results (degrees centigrade)
  Body Temperature measurement results (degrees centigrade)
Patient Measurements (Life Findings, Laboratory Values) | Day one respiratory rate measurement results (.../dak)
  Respiratory rate measurement results (.../dak)
Patient Measurements (Life Findings, Laboratory Values) | Fourth day respiratory rate measurement results (.../dak)
  Respiratory rate measurement results (.../dak)
Patient Measurements (Life Findings, Laboratory Values) | Seventh day respiratory rate measurement results (.../dak)
  Respiratory rate measurement results (.../dak)
Patient Measurements (Life Findings, Laboratory Values) | Fourteenth day respiratory rate measurement results (.../dak)
  Respiratory rate measurement results (.../dak)
Patient Measurements (Life Findings, Laboratory Values) | Twenty-first day respiratory rate measurement results (.../dak)
  Respiratory rate measurement results (.../dak)
Patient Measurements (Life Findings, Laboratory Values) | Day one pulse measurement results (.../dak)
  Pulse measurement results (.../dak)
Patient Measurements (Life Findings, Laboratory Values) | Fourth day pulse measurement results (.../dak)
  Pulse measurement results (.../dak)
Patient Measurements (Life Findings, Laboratory Values) | Seventh day pulse measurement results (.../dak)
  Pulse measurement results (.../dak)
Patient Measurements (Life Findings, Laboratory Values) | Fourteenth day pulse measurement results (.../dak)
  Pulse measurement results (.../dak)
Patient Measurements (Life Findings, Laboratory Values) | Twenty-first day pulse measurement results (.../dak)
  Pulse measurement results (.../dak)
Patient Measurements (Life Findings, Laboratory Values) | Day one blood plessure measurement results (mmHg)
  Blood Plessure measurement results (mmHg)
Patient Measurements (Life Findings, Laboratory Values) | Fourth day blood plessure measurement results (mmHg)
  Blood Plessure measurement results (mmHg)
Patient Measurements (Life Findings, Laboratory Values) | Seventh day blood plessure measurement results (mmHg)
  Blood Plessure measurement results (mmHg)
Patient Measurements (Life Findings, Laboratory Values) | Fourteenth day blood plessure measurement results (mmHg)
  Blood Plessure measurement results (mmHg)
Patient Measurements (Life Findings, Laboratory Values) | Twenty-first day blood plessure measurement results (mmHg)
  Blood Plessure measurement results (mmHg)
Aloe Vera and Propolis Applied Experimental Group and Control Group, Bates-Jensen Wound Assessment Tool Scores | Score change results between day one and day twenty
  Aloe Vera and Propolis Applied Experimental Group and Control Group, Bates-Jensen Wound Assessment Tool Scores
Aloe Vera and Propolis Applied Experimental Group and Control Group, Braden Pressure Injury Risk Scale Assessment Scores | Score change results between day one and day twenty
  Aloe Vera and Propolis Applied Experimental Group and Control Group, Braden Pressure Injury Risk Scale Assessment Scores
Pressure Wound Recovery Time(Day) | It will be recorded on which day the wound healed within three weeks.
  Pressure Wound Recovery Time(Day)
The date the wound culture was taken | For up to three weeks, deep tissue wound culture results will be recorded as (day/month/year).
  It will be recorded as the date (day / month / year) of the wound culture.
Wound culture results | Culture results for three weeks will be recorded.
  The infectious agent growing in the wound culture (Deep tissue culture) will be recorded.
Socio-demographic characteristics of the patient | Sociodemographic characteristics of patients will be recorded for up to three weeks.
  Socio-demographic characteristics of the patient
Patient health history | This outcome measure includes the patient's health history of existing chronic diseases and any co-morbidities developed during the three-week study period.
  Patient health history
Height, Weight | This outcome measure will be used to calculate the patient's body mass index by recording the three-week height and weight measurement results and weight changes over the study period.
  Height .... cm or Weight .... kg
Body Mass İndeks | This outcome measure will be used to calculate the patient's body mass index by recording the three-week height and weight measurement results and weight changes over the study period.
  kg/m2
Current disease information and medications used | This outcome measure includes the patient's current chronic disease-related health history, medications used and any comorbidities developed during the three-week study period, and information on medications used during that three-week period.
  Current disease information and medications used

CONTACTS AND LOCATIONS:
Locations (4):
- Turkey (Türkiye) (4):
  - Haydarpasa Numune Training and Research Hospital, Üsküdar, Istanbul
  - Haydarpasa Numune Training and Research Hospital, Istanbul
  - Bahcelievler State Hospital, Istanbul
  - Medipol Üniversity, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avijgan M, Kamran A, Abedini A. Effectiveness of Aloe Vera Gel in Chronic Ulcers in Comparison with Conventional Treatments. Iran J Med Sci. 2016 May;41(3 Suppl):S30. PMID 27840496
- [Background] Pereira RF, Bartolo PJ. Traditional Therapies for Skin Wound Healing. Adv Wound Care (New Rochelle). 2016 May 1;5(5):208-229. doi: 10.1089/wound.2013.0506. PMID 27134765
- [Background] Khorasani G, Ahmadi A, Hosseinimehr SJ, Ahmadi A, Taheri A, Fathi H. The Effects of Aloe Vera Cream on Split-thickness Skin Graft Donor Site Management: A Randomized, Blinded, Placebo-controlled Study . Wounds. 2011 Feb;23(2):44-8. PMID 25881055
- [Background] Singh S, Gupta A, Gupta B. Scar free healing mediated by the release of aloe vera and manuka honey from dextran bionanocomposite wound dressings. Int J Biol Macromol. 2018 Dec;120(Pt B):1581-1590. doi: 10.1016/j.ijbiomac.2018.09.124. Epub 2018 Sep 21. PMID 30248422
- [Background] Medellin-Luna MF, Castaneda-Delgado JE, Martinez-Balderas VY, Cervantes-Villagrana AR. Medicinal Plant Extracts and Their Use As Wound Closure Inducing Agents. J Med Food. 2019 May;22(5):435-443. doi: 10.1089/jmf.2018.0145. Epub 2019 Apr 3. PMID 30942656
- See also: 2 — https://www.epuap.org/
- See also: 5 — https://doi.org/10.3166/phyto-2018-0075